CLINICAL TRIAL: NCT00696111
Title: PCOS, Sleep Apnea and Metabolic Risk in Women
Brief Title: Metabolic Study of Women With Polycystic Ovary Syndrome and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15872B; 1P50HD057796 (NIH)
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome; Obstructive Sleep Apnea
Keywords: PCOS; OSA; Metabolism; Diabetes
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sleep Apnea, Obstructive; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Depot Lupron and estrogen plus placebo (Experimental): Randomized to receive depot Lupron for 6 weeks. Then randomized again to receive estrogen plus placebo for another 6 weeks.
  Interventions: Drug: Depot Lupron followed by estrogen plus placebo

INTERVENTIONS:
Drug: Depot Lupron followed by estrogen plus placebo — A single intramuscular dose of depot lupron (11.25 mg). Six weeks after injection, subjects will receive daily oral doses of estrogen (2mg) plus placebo for six weeks.
  Other Names: Arm 1

SUMMARY:
The purpose of this study is to look at the metabolic (use of energy) and hormonal features of sleep problems in women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
The prevalence of obesity and chronic sleep loss are at record levels among Americans and evidence continues to emerge to support a causal link between the two conditions. Metabolic abnormalities related to sleep disruption are particularly evident in individuals with obstructive sleep apnea (OSA), a disorder traditionally associated with male gender. While more prevalent in men, OSA is underrecognized in women in part because its clinical and polysomnographic features differ from those of men. Women with polycystic ovary syndrome (PCOS) are particularly susceptible to OSA with at least a 5-fold higher risk for its development compared to obese women without PCOS. This study will enroll obese women with PCOS, with and without OSA. Those with OSA will be randomized to receive CPAP or to receive depot leuprolide to suppress ovarian steroid output over 12 weeks, reassessed at 6 weeks, and then randomized (double-blind, placebo controlled) to 6 weeks of either micronized estrogen + placebo or micronized progestin + placebo. The independent effects of androgen, estrogen, and progesterone on OSA and metabolic function will be assessed. In addition, primary human adipocytes will be prepared from fat biopsies obtained from subjects. Insulin sensitivity will be determined by phospho-specific immunoblotting in conjunction with glucose uptake and anti-lipolysis assays. In parallel, adipocytes from these subjects will be cultured for 1-5 days prior to metabolic assays to ascertain if removal of from circulating factors will improve insulin signaling, or if insulin resistance persists in vitro. Finally, there will be an interface with the Metabolomics Laboratory at Duke University (C. Newgard, Lab Director), and metabolomics assessment will be done on blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS
* Obese (BMI of at least 30 kg/m2)

Exclusion Criteria:

* Diagnosis of nonclassic 21-hydroxylase deficiency, Cushing syndrome, hypothyroidism, or significant elevations in prolactin
* Taking steroid preparations (including oral contraceptives), medications known to alter insulin secretion and/or action, or medications known to influence sleep during the 2 months prior to starting the study
* Positive pregnancy test
* Diagnosis of diabetes mellitus
* Hypertension (systolic > 140 mmHg and/or diastolic > 90 mmhg) not well-controlled on stable medication with either ACE inhibitors or diuretics
* Habitual alcohol use
* Excessive caffeine intake of more than 300 mg/day
* Known peanut allergies, or allergies to medications used in the study
* Hemoglobin < 11g/dL and/or hematocrit < 33%
* Systemic illnesses, including heart, renal, liver, or malignant disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Ehrmann, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Department of Medicine, Section of Endocrinology, Diabetes & Metabolism, Chicago, Illinois, United States

REFERENCES:
- [Background] Hoffman LK, Ehrmann DA. Cardiometabolic features of polycystic ovary syndrome. Nat Clin Pract Endocrinol Metab. 2008 Apr;4(4):215-22. doi: 10.1038/ncpendmet0755. Epub 2008 Feb 5. PMID 18250636
- [Background] Tasali E, Leproult R, Ehrmann DA, Van Cauter E. Slow-wave sleep and the risk of type 2 diabetes in humans. Proc Natl Acad Sci U S A. 2008 Jan 22;105(3):1044-9. doi: 10.1073/pnas.0706446105. Epub 2008 Jan 2. PMID 18172212
- [Background] Dronavalli S, Ehrmann DA. Pharmacologic therapy of polycystic ovary syndrome. Clin Obstet Gynecol. 2007 Mar;50(1):244-54. doi: 10.1097/GRF.0b013e31802f35a0. PMID 17304039
- [Background] Ehrmann DA, Liljenquist DR, Kasza K, Azziz R, Legro RS, Ghazzi MN; PCOS/Troglitazone Study Group. Prevalence and predictors of the metabolic syndrome in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Jan;91(1):48-53. doi: 10.1210/jc.2005-1329. Epub 2005 Oct 25. PMID 16249284
- [Background] Tasali E, Van Cauter E, Ehrmann DA. Relationships between sleep disordered breathing and glucose metabolism in polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Jan;91(1):36-42. doi: 10.1210/jc.2005-1084. Epub 2005 Oct 11. PMID 16219719
- [Derived] Tasali E, Chapotot F, Leproult R, Whitmore H, Ehrmann DA. Treatment of obstructive sleep apnea improves cardiometabolic function in young obese women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Feb;96(2):365-74. doi: 10.1210/jc.2010-1187. Epub 2010 Dec 1. PMID 21123449
- See also: University of Chicago Center for Polycystic Ovary Syndrome — https://www.uchicagomedicine.org/conditions-services/endocrinology-metabolic-disorders/polycystic-ovary-syndrome

RESULTS

PARTICIPANT FLOW:
Groups:
- Specific Aim 1: Baseline analysis comparing PCOS women with OSA to PCOS women without OSA.
Period: Overall Study
Arm/Group | Specific Aim 1
Started | 18
Randomized to Receive Depot Lupron for 6 Weeks | 18
Randomized to Receive Progesterone Plus Placebo for 6 Weeks | 0
Randomized to Receive Continuous Positive Airway Pressure for 6 Weeks | 1
Completed | 1
Not Completed | 17
Not completed — Withdrawal by Subject | 17

BASELINE CHARACTERISTICS:
Arm/Group | Specific Aim 1
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 8
  Caucasian | 9
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Estrogen Levels
Description: Estrogen levels measured every 20 minutes for 24 hours and the the average of those values are presented. The units of measurement are picograms per milliter (pg/ml).
Time Frame: Baseline
Population: The number of patients in Specific Aim 2 is zero, since the one patient randomized to Lupron dropped out.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Specific Aim 1: Women Without Obstructive Sleep Apnea: PCOS women without Obstructive Sleep Apnea
- Specific Aim 1: Women With Obstructive Sleep Apnea: PCOS women with Obstructive Sleep Apnea
- Specific Aim 2: Randomized to receive depot Lupron for 6 weeks. Then randomized again to receive EITHER esgrogen plus placebo OR progesterone plus placebo for another 6 weeks.
  Depot Lupron followed by estrogen plus placebo.: A single intramuscular dose of depot lupron (11.25 mg). Six weeks after injection, subjects will receive daily oral doses of estrogen (2mg) plus placebo for six weeks.
  Depot Lupron followed by progesterone plus placebo.: A single intramuscular dose of depot lupron (11.25 mg). Six weeks after injection, subjects will receive daily oral doses of progesterone (200mg) plus placebo for six weeks.
- Specific Aim 3: Randomized to receive CPAP (continuous positive airway pressure) treatment for 6 weeks.
  CPAP: CPAP (continuous positive airway pressure) treatment at home for six weeks.
Arm/Group | Specific Aim 1: Women Without Obstructive Sleep Apnea | Specific Aim 1: Women With Obstructive Sleep Apnea | Specific Aim 2 | Specific Aim 3
Number analyzed (Participants) | 13 | 5 | 0 | 1
pg/ml | 73.3 (32.5) | 69.9 (14.1) |  | 61.0 (18.2)

2. Primary Outcome: Sleep Efficiency Measured at Baseline
Description: Sleep efficiency recorded with polysomnography minimum value = 0%, maximum value = 100%, higher values are a better outcome.
Time Frame: Baseline
Population: Patients dropped out after randomization.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Specific Aim 1: Women Without OSA: PCOS women without Obstructive Sleep Apnea.
Arm/Group | Specific Aim 1: Women Without OSA | Specific Aim 1: Women With Obstructive Sleep Apnea | Specific Aim 2 | Specific Aim 3
Number analyzed (Participants) | 13 | 5 | 0 | 1
Percentage | 93.2 (4.0) | 86.7 (7.0) |  | 92.3

3. Primary Outcome: Total Testosterone
Description: Total Testosterone levels measured every 20 minutes for 24 hours and the average of those values are presented. The units of measurement are picograms per milliter (pg/ml).
Time Frame: Baseline
Population: patients dropped out after randomization
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Specific Aim 1: Women Without Obstructive Sleep Apnea | Specific Aim 1: Women With Obstructive Sleep Apnea | Specific Aim 2 | Specific Aim 3
Number analyzed (Participants) | 13 | 5 | 0 | 1
pg/ml | 70.5 (44.7) | 50.9 (26.4) |  | 45.3 (14.8)

4. Secondary Outcome: Intravenous Glucose Tolerance Test
Description: Acute Insulin Response measured by the intravenous glucose tolerance test measured during baseline. The unit of measurement is mg/dl.
Time Frame: Baseline
Population: Patients dropped out after randomization
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Specific Aim 1:PCOS Women Without Obstructive Sleep Apnea: Women without Obstructive Sleep Apnea.
- Specific Aim:1 PCOS Women With Obstructive Sleep Apnea: Women with Obstructive Sleep Apnea
- Specific Aim3: Randomized to receive CPAP (continuous positive airway pressure) treatment for 6 weeks.
  CPAP: CPAP (continuous positive airway pressure) treatment at home for six weeks.
Arm/Group | Specific Aim 1:PCOS Women Without Obstructive Sleep Apnea | Specific Aim:1 PCOS Women With Obstructive Sleep Apnea | Specific Aim 2 | Specific Aim3
Number analyzed (Participants) | 13 | 5 | 0 | 1
mg/dl | 938.5 (770.1) | 730.6 (478.1) |  | 189.5

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the baseline analysis 12 days for patients in Aim 1. For participants randomized to CPAP treatment (Aim 3), adverse events were monitored during the 6 weeks of CPAP treatment.
Description: Adverse events
Arm/Group | Specific Aim 1 | Specific Aim 2 | Specific Aim 3
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/18 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT00696111/Prot_SAP_000.pdf